CLINICAL TRIAL: NCT01292694
Title: Contribution of Angiotensin II to Supine Hypertension in Autonomic Failure
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Could not enroll enough participants, and lost funding.
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor and Associate Director Clinical Research Center, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 101618
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Hypertension; Pure Autonomic Failure; Multiple System Atrophy
Keywords: supine hypertension; autonomic failure; angiotensin; losartan; captopril
MeSH Terms: conditions — Hypertension; Pure Autonomic Failure; Multiple System Atrophy | interventions — Losartan; Captopril

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Losartan (Experimental): Angiotensin II AT1 receptor antagonist which blocks the actions of angiotensin II
  Interventions: Drug: Losartan
- Captopril (Experimental): ACE inhibitor which blocks the formation of angiotensin II
  Interventions: Drug: Captopril
- Placebo Tablet (Placebo Comparator): A placebo tablet will be provided by the Vanderbilt Investigational Drug Service for these studies.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan — Oral, single-dose, 50 mg tablet
  Other Names: Cozaar
  Arms: Losartan
Drug: Captopril — Oral, single-dose, 50 mg tablet
  Other Names: Capoten
  Arms: Captopril
Drug: Placebo — Oral, single administration, gelatin capsule filled with microcrystalline cellulose
  Arms: Placebo Tablet

SUMMARY:
The purpose of this study is to test the hypothesis that angiotensin II plays a role in the supine hypertension of primary autonomic failure. To determine the contribution of angiotensin II to renin and blood pressure regulation in autonomic failure, patients with multiple system atrophy [MSA] or pure autonomic failure [PAF] and supine hypertension will undergo medication testing with the angiotensin II receptor blocker losartan. The investigators will compare the biochemical and hemodynamic effects between MSA and PAF patients. In a subset of patients, the investigators will also give the ACE inhibitor captopril. Our primary endpoint will be changes in plasma renin activity, and subsequent components of the circulating renin-angiotensin system, in response to angiotensin II blockade. Our secondary outcome will be changes in hemodynamic measures during administration of these drugs.

DETAILED DESCRIPTION:
Primary autonomic failure is a disabling condition characterized by orthostatic hypotension. It is less well appreciated that at least 50% of these patients have high blood pressure when lying down [supine hypertension]. The mechanisms underlying supine hypertension in autonomic failure remain poorly understood. The hypertension in MSA patients may be explained by residual sympathetic tone, possibly acting on hypersensitive adrenoreceptors and unrestrained by the lack of baroreflex modulation. In contrast, the hypertension in PAF is associated with increased vascular resistance in the absence of residual sympathetic tone. However, the factors driving an elevation in either sympathetic or vascular tone in these patients remain unclear.

The investigators hypothesize that angiotensin II, a hormone widely implicated in blood pressure regulation, plays a role in the supine hypertension of autonomic failure. To determine the contribution of angiotensin II to renin and blood pressure regulation in autonomic failure, the investigators will administer the angiotensin II receptor blocker losartan to MSA and PAF patients with supine hypertension. The primary endpoint will be changes in plasma renin activity, and subsequent components of the circulating renin-angiotensin system, in response to angiotensin II blockade. The secondary outcomes will be the decrease in blood pressure and changes in heart rate, cardiac output, stroke volume and systemic vascular resistance during administration of these drugs.

Subjects will be studied on 2 separate days, one with oral administration of placebo and the other with losartan [50 mg]. The order of administration will be randomized in a single-blind manner. The investigators will collect blood samples before and every 2 hours after administration for up to 6 hours to determine if angiotensin II regulates plasma renin activity, and other components of the circulating renin-angiotensin system, in autonomic failure. The investigators will also obtain hemodynamic measurements before and every 1 hour (blood pressure and heart rate) or 2 hours (cardiac output, stroke volume and systemic vascular resistance) after drug administration.

In a subset of patients the investigators will also administer the ACE inhibitor captopril [50 mg] on a separate study day using the same methods. Captopril is less specific for assessing the role of angiotensin II to hypertension. However, it may provide important information on the mechanism for angiotensin II formation in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with autonomic failure who exhibit supine hypertension and are in the hospital already participating in the study "The Evaluation and Treatment of Autonomic Failure [IRB # 000814]
* Supine hypertension, defined as systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 90 mm Hg
* Males and females of all races, between 18 to 85 years of age
* Able and willing to provide informed consent with the understanding that they may withdraw consent at any time without prejudice to future medical care

Exclusion Criteria:

* All medical students
* Pregnant women
* Patients with a history of angioedema
* Patients with a known allergy to any ACE inhibitor or angiotensin receptor blocker
* High-risk patients [e.g. heart failure, symptomatic coronary artery disease, liver impairment, history of stroke or myocardial infarction]
* Patients with hemoglobin < 10.5 [or hematocrit < 32]
* Inability to give, or withdraw, informed consent
* Other factors which in the investigator's opinion would prevent the patient from completing the protocol including clinically significant abnormalities in clinical, mental or laboratory testing

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Changes in plasma renin activity and subsequent components of the circulating renin-angiotensin system | 0 - 6 hours post administration
  Changes in supine plasma renin activity and aldosterone following drug administration

SECONDARY OUTCOMES:
Changes in blood pressure | 0 - 6 hours post administration
  Changes in supine blood pressure following drug administration
Changes in heart rate, cardiac output, stroke volume and systemic vascular resistance | 0 - 6 hours post administration
  Changes in supine systemic hemodynamics following drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States